CLINICAL TRIAL: NCT03436537
Title: Development and Validation of the Periodontal Aesthetic Perception Scale in Patients With Periodontal Problems
Status: Completed | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Ozge Gokturk, asst. assoc., Tokat Gaziosmanpasa University
Other Study IDs: 17-KAEK-131
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Gingival Enlargement; Gingival Recession
Keywords: aesthetic; development; periodontal; reliability; validity
MeSH Terms: conditions — Gingival Hyperplasia; Gingival Recession

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Gingival recession (GR) group: GR group answered the self-reported 7-item questionnaire for Periodontal aesthetic perception scale
  Interventions: Other: Periodontal Aesthetic Perception Scale
- Gingival enlargement (GE) group: GE group answered the self-reported 7-item questionnaire for Periodontal aesthetic perception scale.
  Interventions: Other: Periodontal Aesthetic Perception Scale
- periodontal healthy (H) group: H group answered the self-reported 7-item questionnaire for Periodontal aesthetic perception scale.
  Interventions: Other: Periodontal Aesthetic Perception Scale

INTERVENTIONS:
Other: Periodontal Aesthetic Perception Scale — Patients answered the self-reported 7-item questionnaire for Periodontal aesthetic perception scale

SUMMARY:
Aesthetics for individuals become increasingly important, while the aesthetic effects of periodontal disease is an important issue that should be assessed by the patient's perception.

The results demonstrate that the periodontal aesthetic perception scale showed reliable and valid scores in healthy controls and periodontal patients.

The periodontal aesthetic perception scale may be an appropriate tool to assess periodontal esthetic in clinical and research settings.

DETAILED DESCRIPTION:
Aim: The aim of this study is to develop and validate a periodontal aesthetic specific tool to assess aesthetic conditions perceived by patients with periodontal problems.

Methods: With patient interviews were identified a total of 22 statements that describe the non-aesthetic gingival appearance. These 22 items were reviewed by the dentists and then Periodontologists and the number of items in the survey was reduced to 7. Subsequently, three groups of patients were included in the study: Gingival recession (GR) group, gingival enlargement (GE) group and periodontal healthy (H) group. Consequently, the validity and reliability of the periodontal aesthetic perception scale (PAPS) were examined.

Results: According to the results of the Exploratory Factor Analysis (EFA), 1 item was removed from the scale. The final 6-item questionnaire was shown to have a two-domain structure. Cronbach's alpha for the whole scale was .766. The interclass correlation coefficients (ICCs) values were between 0.98 and 1.00, demonstrating excellent agreement. Overall, these findings indicated that the PAPS has good reliability.

Conclusion: This reliable, valid and short questionnaire specific to aesthetic conditions perceived by patients with periodontal problems may serve as a valued instrument in future clinical trials.

ELIGIBILITY:
Inclusion criteria for gingival recession group:

- The presence of gingival recession (Miller Class I, II, III, or IV) in maxillary and mandibular anterior teeth.

Inclusion criteria for gingival enlargement group:

-The presence of gingival enlargement (Grade 0, I, II, III, or IV) in maxillary and mandibular anterior teeth.

Exclusion Criteria for all groups:

* The presence of prosthesis, tooth loss or caries in the anterior teeth
* The precence of the psychological or systemic disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who fulfilled the criteria for inclusion presenting at the periodontology clinic were asked to participate in the study and those agreeing to interview were asked how and what aesthetically disturbing symptoms in their gingiva.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Validity of PAPS | 6 months
  The KMO (Kaiser-Meyer-Olkin) test produced a value of 0.80, which was greater than the recommended threshold value of 0.50.

CONTACTS AND LOCATIONS:
Overall Officials: Ozge Gokturk, Study Director — Study Principal Investigator
Locations (1):
- Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Result] Slade GD, Spencer AJ. Development and evaluation of the Oral Health Impact Profile. Community Dent Health. 1994 Mar;11(1):3-11. PMID 8193981